CLINICAL TRIAL: NCT01556399
Title: A Correlation of the Endoscopic Characteristics of Duodenal and Ampullary Laterally Spreading Tumours With Their Somatic or Germline Mutations.
Brief Title: Endoscopic Characteristics of Duodenal and Ampullary Lesions
Acronym: DUO/AMP-LST
Status: Completed | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: LST-UGIM
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Duodenal Diseases
Keywords: Duodenal adenoma; Ampullary adenoma
MeSH Terms: conditions — Duodenal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adenoma tissue sample and control "regular" tissue sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Duodenal adenomas: Patients who consent to participate in this study will have a small sample of their adenoma and normal tissue sent for molecular testing.
  Interventions: Other: Tissue Sampling

INTERVENTIONS:
Other: Tissue Sampling — A small sample of the duodenal adenoma will be obtained for molecular testing. The remaining adenoma will be sent for regular histological testing.

SUMMARY:
The purpose is to investigate whether polyps that look different at endoscopy, have formed via different mutations and have different risks of turning into cancer.

DETAILED DESCRIPTION:
Laterally spreading tumours (LSTs), are polyps that have a lateral extension along the duodenal wall with minimal vertical growth. It has become evident over the last few years that rather than being a single entity requiring an accumulation of mutations, Duodenal and ampullary cancer is in fact a heterogenous disease forming via multiple distinct genetic pathways. It is therefore hypothesised that different polyp types have different genetic abnormalities, and potentially form via distinct genetic pathways, although this theory has not been widely examined.

This knowledge would be important in furthering our understanding of the development of cancer. There is accumulating evidence that genetic abnormalities may be a better predictor of cancer behaviour than histological grade. Additionally, guidelines for endoscopy surveillance are currently a one size fits all approach that do not reflect the genetic heterogeneity of the disease and the knowledge that only 5% of polyps progress to cancer. Genetic studies may assess future cancer risk to a person in polyps once removed and plan surveillance endoscopy frequency.

ELIGIBILITY:
Inclusion Criteria:

* Intention to perform Endoscopic Mucosal Resection
* Adenoma equal to or greater than 20mm
* over 18 years of age
* Able to give informed consent to involvement in trial

Exclusion Criteria:

* Pregnancy
* Lactation: currently breastfeeding
* Taken clopidogrel within 7 days
* Taken warfarin within 5 days
* Had full therapeutic dose unfractionated heparin within 6 hours
* Had full therapeutic dose low molecular weight heparin (LMWH) within 12 hours
* Known clotting disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Duodenal and/or ampullary adenomas or cancers.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-11; Primary Completion 2017-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Significant differences in molecular abnormalities. | Specimens will be stored and used for up to 15 years
  The aim of this project is to look for statistically significant differences in molecular abnormalities from the three known genetic pathways, between the two different morphological types, granular and non-granular, to potentially demonstrate that these different polyps form via different genetic pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, FRACP, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia